CLINICAL TRIAL: NCT05405348
Title: The Effect of Food Intake During Hemodialysis on Blood Pressure: A Non-randomized Experimental Trial
Brief Title: The Effect of Food Intake During Hemodialysis on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: melek avcı (Other)
Responsible Party: Sponsor-Investigator, melek avcı, Department of Internal Medicine Nursing, MsC, RN, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-KAEK-20-547
Record Dates: First submitted 2022-03-23; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Renal Dialysis
Keywords: hemodialysis; blood pressure; intradialytic food intake; intradialytic hypotension
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: In this study, one group patients were observed two different times. First meeting(T0, patients took routine care which include fed state during the hemodialisis.Second meeting (T1) patients took intervention which include fasting state during the hemodialisis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group received routine care (T0)
- Intervention (Experimental): Same patients, one week after T0, T1 was applied in middialysis. In T1, patients did not consume food at least half an hour before coming to hemodialysis. They also did not consume any food during hemodialysis.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The patients did not eat anything during hemodialysis.
  Arms: Intervention

SUMMARY:
Intradialytic hypotension is one of the most common complications associated with food intake during hemodialysis. Whether patients should be allowed to eat during hemodialysis is still a moot point.

This nonrandomized experimental trial investigated the effect of food intake during hemodialysis on blood pressure of patients. The sample consisted of 54 chronic patients receiving hemodialysis treatment. Researchers monitored the patients in two hemodialysis sessions; first meeting (T0) and second meeting (T1) which is one week later from T0. In the first meeting which is ''hemodialysis in fed state'', they ate the standard food served by the clinic at regular hours which means routine care of hemodialysis clinic. In the second meeting which is ''hemodilaysis in fasting state'', they did not eat anything during hemodialysis which means intervention part of the study. Both hemodyalisis in fed and fasting state, researchers recorded patient's blood pressure were monitozied in the mid-hemodiyalsis sessions. Patient' s sociodemographic and disease characteristics were recorded. Patient' s blood pressure monitorized by the ambulatory blood pressure monitor.

DETAILED DESCRIPTION:
Researchers monitored the patients in two hemodialysis sessions; first meeting (T0) and second meeting (T1) which is one week later from T0. In the first meeting which is ''hemodialysis in fed state'', they ate the standard food (in clinic routine) served by the clinic at regular hours which means routine care of hemodialysis clinic. In the second meeting patients did not eat anything during hemodialysis which means intervention part of the study. Both hemodyalisis in fed and fasting state, researchers recorded patient's blood pressure were monitozied in the mid-hemodiyalsis sessions. Patient' s sociodemographic and disease characteristics were recorded. Patient' s blood pressure monitorized by the ambulatory blood pressure monitor.

Blood pressure measurements were made using Suntech Bravo Ambulatory Blood Pressure Monitoring (Morrisville, USA). Blood pressure was evaluated in the supine position with the use of a brachial cuff. The blood pressure measurement was made in the midweek dialysis session on the day of the measurement. Before the patient entered hemodialysis, an ambulatory blood pressure monitor was placed and blood pressure was measured at 15-minute intervals throughout the 4-hour hemodialysis session. A total of 16 measurements were made. The patients did not consume any food during the 4-hour dialysis session.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Having CKD and being in the hemodialysis program
* Having the ability to understand and speak
* Being on HD treatment for 6 months or longer
* Weight gain of 4 kg or less between two HD sessions
* Standard HD is applied 3 days a week for 4 hours

Exclusion Criteria:

* The patient's communication difficulties, speech and understanding deterioration,
* Being on dialysis for less than 6 months,
* Interdialytic weight gain of more than 4kg,
* The patient is not suitable for blood pressure measurement from the arm,
* The patient used antihypertensive before HD,
* Entering HD less than or more than 3 days a week,
* More or less than 4 hours of HD input.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Effect of food consumption on intradialytic blood pressure | 3 month
  Blood pressure measurements were made using Suntech Bravo Ambulatory Blood Pressure Monitoring (Morrisville, USA). Blood pressure was evaluated in the supine position with the use of a brachial cuff. The blood pressure measurement was made in the midweek dialysis session on the day of the measurement. Before the patient entered hemodialysis, an ambulatory blood pressure monitor was placed and blood pressure was measured at 15-minute intervals throughout the 4-hour hemodialysis session. A total of 16 measurements were made.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Avcı, PhD Student, Study Director — Akdeniz University; Fatma Arikan, PhD, RN, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)